CLINICAL TRIAL: NCT05039697
Title: Normobaric Hyperoxia Combined With Endovascular Therapy in Patients With Stroke Within 6 Hours of Onset：Longterm Outcome Analysis
Brief Title: Normobaric Hyperoxia Combined With Endovascular Therapy in Patients With Stroke Within 6 Hours of Onset：Longterm Outcome
Acronym: NBOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPENS-2L
Record Dates: First submitted 2021-04-06; First posted 2021-09-09 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Stroke, Acute; Hypoxia-Ischemia, Brain; ENDOVASCULAR TREATMENT
MeSH Terms: conditions — Stroke; Hypoxia-Ischemia, Brain | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NBO group Normobaric Hyperoxia combined with endovascular mechanical thrombectomy (Experimental): Within 6 hours after stroke onset, patients were randomized into the NBO group and immediately given 100% oxygen inhalation (no more than 30minutes after admission) at a ventilation rate of 10L/min using a sealed non-ventilating oxygen storagemask and keep giving oxygen for 4 hours. If the patient needs to be intubated with a ventilator to maintain ventilation, the FiO2 should be set to 1.0.
  Interventions: Other: oxygen
- Control group Inhale air placebo plus endovascular mechanical thrombectomy (Placebo Comparator): For Sham NBO group, Patients were immediately given oxygen inhalation (no more than 30 minutes after admission) at a ventilation rate of 1l/min using the same mask and keep giving oxygen for 4 hours. If the patient needs to be intubated with a ventilator to maintain, the FiO2 should be set to 0.3 and gradualy incerased if spO2≤94%
  Interventions: Other: oxygen

INTERVENTIONS:
Other: oxygen — deliver high flow oxygen (10L/min)

SUMMARY:
The overall incidence of good outcome for AIS following endovascular treatment is only proximately 50%. Whether NBO was safe and effective to improve acute ischemic stroke prognosis is still unclear. The investigators' hypothesis is thatNBO is a safe and effective strategy to improve longterm outcome in AIS patients undergoing endovascular treatment.

DETAILED DESCRIPTION:
NBO therapy is to deliver high flow oxygen (10L/min) through an oxygen storage mask. This treatment should be started in the emergency room immediately after the patient is randomized into the group, and oxygen should be continued for 4 hours.

In previous clinical studies of NBO, patients who have not receive revascularization often choose NBO for 8 hours, and studies have concluded that oxygen inhalation for more than 10 hours may bring about the risk of oxygen poisoning. However, a too short treatment time may not bring benefits. Secondly, ideally, we want to ensure that stroke patients receive NBO treatment before achieving reperfusion to protect the ischemic brain tissue, and add 1-2 hours after reperfusion. In the clinical environment after the patient arrives in the emergency department, it takes 2-3 hours to complete the revascularization process. Therefore, we believe that 4 hours of oxygen inhalation is reasonable. And our single-center study also supports that NBO treatment for 4 hours is beneficial.

The specific content is as follows: In the emergency room, patients who are assessed for suspected large blood vessels of acute anterior circulation will be randomized after signing the informed consent. If the subject is randomly divided into NBO+ET group, by putting the patient on Oxygen mask, and then immediately give oxygen (10L/min). NBO treatment is no later than half an hour after randomization. Oxygen comes from the hospital's oxygen center and is transported through wall pipes (oxygen concentration: 100%). The oxygen mask and the wall oxygen are connected by a 1.5 meter long oxygen pipe. When the patient is transferred to the operating room, we provide oxygen through a portable oxygen cylinder (capacity: 4L). In addition, in the operating room and intensive care unit, patients continue to be given wall oxygen therapy until the oxygen inhalation lasts for 4 hours. The arterial blood gas was drawn after 4 hours of oxygen inhalation. The control group directly inhales room air through the patient's nasal cavity without using any equipment. At the same time, patients in the control group were also drawn blood gas analysis at corresponding time points (approximately 4 hours after randomization).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* The clinical symptoms and signs are consistent with acute anterior circulation large vessel occlusion;
* NIHSS score ≥ 10 points;
* (Level of consciousness) NIHSS score 0 or 1;
* The time from onset to randomization is within 6 hours of onset;
* The mRS score before stroke is 0-1;
* The patient has good compliance and can complete the operation with local anesthesia;
* The patient can cooperate with this study and follow-up in the future
* Patient and family members sign informed consent。-

Exclusion Criteria:

* Rapid neurological function improvement, NIHSS score less than 10 points, or evidence of vessel recanalization prior to randomization;
* Seizures at stroke onset;
* Intracranial hemorrhage;
* Symptoms suggestive of subarachnoid hemorrhage, even if CT scan was normal;
* Platelet count of less than 100,000 per cubic millimeter;
* Severe hepatic or renal dysfunction;
* Active and chronic obstructive pulmonary disease or acute respiratory distress syndrome;
* >3 L/min oxygen required to maintain peripheral arterial oxygen saturation (SaO2) 95% as per current stroke management guidelines;
* Medically unstable;
* Life expectancy<90 days;
* Evidence of intracranial tumor;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2024-02-04 (Actual); Study Completion 2024-02-04 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale | 1 year ± 30 days after randomization
  the mRs is an ordinal disability score of 7 categories (0=no symptoms to 5=severe disability,and 6=death)

SECONDARY OUTCOMES:
EuroQol- 5 Dimension (EQ-5D) | 1 year ± 30 days after randomization
  EuroQol five dimensions questionnaire (EQ-5D)EQ-5D is an instrument which evaluates the generic quality of life developed in Europe and widely used. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
The proportion of good prognosis | 1 year ± 30 days after randomization
  the mRs is an ordinal disability score of 7 categories (0 = no symptoms to 5 = severe disability, and 6 = death);The ratio of 0 to 2
Functional independence | 1 year ± 30 days after randomization
  The Proportion of mRS 0-1
The Proportion of mRS 0-3 | 1 year ± 30 days after randomization
  secondary clinical efficacy endpoint
Barthel Index (BI) | 1 year ± 30 days after randomization
  he BI is an ordinal disability score of 10 categories(range from 0 to 100, higher values indicate better prognosis);
All-cause mortality | 1 year ± 30 days after randomization
  clinical safety endpoint;
New major vascular events | 1 year ± 30 days after randomization
  clinical safety endpoint; Major vascular events include fatal or nonfatal cardiac events, fatal or nonfatal stroke, or fatal or nonfatal major peripheral arterial or thrombo-embolic events.
kaplan-meier curve | 1 year ± 30 days after randomization
  clinical efficacy endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD, Study Chair — Xuan Wu Hospital#Capital Medical University
Locations (1):
- Baojun Hou, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei M, Wang X, Wang S, Liu S, Ji X, Li W. Protocol for a prospective 1-year follow-up investigation on normobaric hyperoxia in conjunction with endovascular treatment for acute ischemic stroke (OPENS-2L) trial. Brain Circ. 2025 Mar 31;11(2):127-134. doi: 10.4103/bc.bc_29_24. eCollection 2025 Apr-Jun. PMID 40520063